CLINICAL TRIAL: NCT05581316
Title: An Investigation of the Effect of Types of Catheters on Bloodstream Infection in Patients With Major Burns: Prediction With Procalcitonin and Prognosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hasan Kalyoncu University (Other)
Responsible Party: Principal Investigator, Murat Ali ÇINAR, assistive professor, Hasan Kalyoncu University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: MAC2022-N
Record Dates: First submitted 2022-10-11; First posted 2022-10-14 (Actual); Last update posted 2022-10-14 (Actual); Status verified 2022-10

CONDITIONS: Burns
Keywords: burns; Blood stream infections; procalcitonin
MeSH Terms: conditions — Burns | interventions — Platelet Count

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- patients who use peripheral venous catheters (Experimental): Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center. The above examinations at the Laboratories of the December 25th State Hospital, Ministry of Health of the Republic of Turkey, were retrieved retrospectively from the hospital database
  Interventions: Diagnostic Test: Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center.
- patients who use venous catheters (Experimental): Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center. The above examinations at the Laboratories of the December 25th State Hospital, Ministry of Health of the Republic of Turkey, were retrieved retrospectively from the hospital database
  Interventions: Diagnostic Test: Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center.

INTERVENTIONS:
Diagnostic Test: Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center. — This patients who were included in this study were assessed for four weeks from the first day of hospitalization and taken to the treatment program. All patients who use peripheral venous catheters in this group.

SUMMARY:
Bloodstream infections and catheter-related infections frequently occur in burn patients. It is important to correctly assess and manage these infections. The present study aimed to investigate the effects of catheter types used in major burn patients on bloodstream infections as well as to predict sepsis status and manage its prognosis using a procalcitonin biomarker.

DETAILED DESCRIPTION:
Aim:

Bloodstream infections and catheter-related infections frequently occur in burn patients. It is important to correctly assess and manage these infections. The present study aimed to investigate the effects of catheter types used in major burn patients on bloodstream infections as well as to predict sepsis status and manage its prognosis using a procalcitonin biomarker.

Materials and Methods:

A total of 34 patients admitted to the intensive care unit of the Burn Center, December 25th State Hospital, Ministry of Health, between 2019 and 2022, were included in the study conducted at the Department of Physiotherapy and Rehabilitation, Faculty of Health Sciences, Hasan Kalyoncu University.

Study inclusion criteria

* Conscious and cooperative (based on the Glasgow coma score; eyes open spontaneously (E): 4, obeys commands (M): 6, oriented verbal (V) response: 5; and E4M6V5);
* Enterally fed, aged over 18 years;
* No antibiotic treatment from hospitalization to discharge;
* Meets the major burn class standards defined by the American Burn Association; and
* Stable hemodynamic values and vital signs with no need for inotropic medication.

Study exclusion criteria

* Organ dysfunctions or multiple organ failures
* Antibiotics treatment Nutrient types and diets were the same in all groups. All patients received similar standard medical care and treatment from the time of emergency admission and acute care of the burn injury until the time of discharge. In addition, types and numbers of clinical interventions, such as surgical debridement and grafting, were similar in all groups. All patients who were included in this study were assessed for four weeks from the first day of hospitalization and taken to the treatment program.

Patients included in the study were divided into two groups based on whether they used PVCs or CVCs. Patients' procalcitonin, thrombocyte, and leukocyte levels were assessed every other day for 4 weeks, beginning on the first day they were admitted to the burn center. The above examinations at the Laboratories of the December 25th State Hospital, Ministry of Health of the Republic of Turkey, were retrieved retrospectively from the hospital database.

.

ELIGIBILITY:
Inclusion Criteria:

* Conscious and cooperative (based on the Glasgow coma score; eyes open spontaneously (E): 4, obeys commands (M): 6, oriented verbal (V) response: 5; and E4M6V5);
* Enterally fed, aged over 18 years;
* No antibiotic treatment from hospitalization to discharge;
* Meets the major burn class standards defined by the American Burn Association; and
* Stable hemodynamic values and vital signs with no need for inotropic medication.

Exclusion Criteria:

* Organ dysfunctions or multiple organ failures • Antibiotics treatment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Level of procalcitonin | Each participant will be evaluated for 4 weeks
  blood test
Level of thrombocyte | Each participant will be evaluated for 4 weeks
  blood test
Level of leukocyte | Each participant will be evaluated for 4 weeks
  blood test

CONTACTS AND LOCATIONS:
Overall Officials: MURAT A ÇINAR, DR, Principal Investigator — Study Principal Investigator
Locations (1):
- Hasan Kalyoncu University, Gaziantep, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Manda T, Nishigaki F, Mori J, Shimomura K. Important role of serotonin in the antitumor effects of recombinant human tumor necrosis factor-alpha in mice. Cancer Res. 1988 Aug 1;48(15):4250-5. PMID 3390820